CLINICAL TRIAL: NCT02060708
Title: Measuring the Stimulated Brain: Determining the Specificity of High Definition Electrical Brain Stimulation Using Simultaneous Magnetoencephalography
Brief Title: Determining the Specificity of High Definition Electrical Brain Stimulation Using Simultaneous Magnetoencephalography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Douglas Cheyne, Senior Scientist and Associate Professor, Diagnostic Imaging, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1000042023
Record Dates: First submitted 2014-02-06; First posted 2014-02-12 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Real HD-tDCS; Sham HD-tDCS; Visual Task; Motor Task; Auditory Task; Working Memory Task

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- Real HD-tDCS first, Sham HD-tDCS second (Other): Real HD-tDCS will be applied in the first session Sham HD-tDCS will be applied in the second session (at least one week after the first session)
  Interventions: Device: HD-tDCS
- Sham HD-tDCS first, Real HD-tDCS second (Other): Sham HD-tDCS will be applied in the first session Real HD-tDCS will be applied in the second session (at least one week after the first session)
  Interventions: Device: HD-tDCS

INTERVENTIONS:
Device: HD-tDCS — HD-tDCS non-invasive brain stimulation using this same device (Soterix) has been designated a 'non-significant risk' by the US FDA.
  Other Names: High Definition Transcranial Direct Current Stimulation

SUMMARY:
Non-invasive human brain stimulation using weak transcranial direct-current stimulation (tDCS) has been thousands of times in research studies over the past fifteen years as a therapy to help improve the effectiveness of repeated training sessions (e.g., hand exercises in the context of daily physiotherapy), due to its safety, tolerability, convenience and cost-effectiveness. tDCS works by temporarily enhancing brain activity during performance of a specific task, helping with learning and training.

The investigators will use magnetoencephalography (MEG) brain imaging to view the real-time effects of high definition (HD) tDCS on several brain areas involved in vision, hearing, movement, and memory. The investigators hypothesize that changing the task (auditory, visual or memory task) but keeping the position of the electrodes over the motor cortex will result in modulation of brain activity in only the central target motor area, and not on non-target temporal, occipital or pre-frontal areas.

ELIGIBILITY:
Inclusion Criteria:

* Normal hearing and vision

Exclusion Criteria:

* Current pregnancy
* Presence of metallic implants in the head
* Use of any medications
* Any history of mental health or neurological conditions
* Inability to perform any of the tasks for any reason

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in brain activity | Immediate (20 minutes)
  Assessment of changes in brain activity will be done using both event-related and frequency domain beam former localization.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada